CLINICAL TRIAL: NCT02658877
Title: In Situ Analysis of Sputum-derived Cellular Targets After Xolair (Omalizumab).
Brief Title: Sputum-derived Cellular Targets After Xolair (Omalizumab)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty recruiting subjects
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-01160
Record Dates: First submitted 2015-12-17; First posted 2016-01-20 (Estimated); Results first posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Asthma
Keywords: Xolair; corticosteroids; asthma; long-acting beta-agonists
MeSH Terms: conditions — Asthma | interventions — Omalizumab; Adrenal Cortex Hormones; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Omalizumab (Experimental)
  Interventions: Drug: Omalizumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omalizumab — Omalizumab will be dosed according to dosing and U.S. administration guidelines for omalizumab. Omalizumab will be dosed every 2-4 weeks based on the patient's pre treatment serum IgE level (IU/mL) and initial visit body weight (kg). Omalizumab will be delivered as a subcutaneous injection. Standard safety precautions for dosing will be observed, including clinical observation after dosing, and provision of an epinephrine pen. Maintenance asthma treatment will remain unchanged.
  Other Names: Xolair; corticosteroids
  Arms: Omalizumab
Drug: Placebo — Saline with a volume of injection frequency indicated based on the patient's serum IgE and body weight, delivered subcutaneously and supplied by Novartis Pharma.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to identify additional mechanisms of action of omalizumab that will lead to improved stratification of patients for treatment. Understanding the response of specific innate immune effector cells in the lung can provide clues to these questions. Investigators will use non-invasive measures of a discrete cell population to examine the downstream effects of omalizumab treatment in the lung. Information derived from these studies will help clarify mechanisms of action of omalizumab and help identify potential tools for patient endotyping and stratification for therapeutic interventions.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double blind, 16-week intervention study to show feasibility and proof of concept. Analysis of whole induced sputum is under development for endotyping for asthma, allowing sampling of rare cells from conducting airways, repeated sampling, and cell-specific detailed genomic evaluation. Investigators have developed a novel technique to simultaneously enrich innate immune cells from sputum. This technique allows for in situ analyses of sputum-derived human bronchial epithelial cells (sHBEC). The non-invasive nature of the technique provides a unique tool for in vivo human studies.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosed asthma
* Lung function (one or more of the following documented in the 5 years before enrollment or demonstration during screening) 1. Bronchial hyper responsiveness (BhR) confirmed by ≥ 12% improvement in FEV1 post bronchodilator within the previous 5 years, or 2. Methacholine PC20 < 16mg/dl within the previous 5 years
* Severity Criteria: Moderate-persistent asthma defined by the American Thoracic Society (ATS)
* Asthma Control: Partly or uncontrolled asthma according to GINA 2012 guidelines (at least three of the following features: daytime symptoms more than 2 times/week, limitation of activities, nocturnal symptoms, need for rescue inhaler > 2 times/week, FEV1 <80% predicted)
* Stable use of moderate-high dose inhaled corticosteroids in previous 3 months (definition derived from GINA 2012 guidelines: e.g. fluticasone propionate >250 mcg/day, budesonide > 400mcg/day)
* Ability to perform induced sputum maneuvers
* Presence of elevated allergen IgE to any perennial aeroallergen

Exclusion Criteria:

* Pulmonary function: FEV1 ≤ 70% predicted
* Any major chronic illness including but not limited to Chronic Obstructive Pulmonary Disease (COPD), uncontrolled hypertension, coronary artery disease, bronchiectasis, congestive heart failure, stroke, cystic fibrosis, insulin-dependent diabetes mellitus, renal failure, liver disorders, immunodeficiency state, or other condition that would interfere with participation in the study
* Current or > 10 pack a year pack-year tobacco use
* Any investigational study within previous 1 month
* Inability to perform baseline measurements
* Inability to contact by telephone
* Pregnancy at screening and failure to use double barrier pregnancy protection in woman of childbearing age
* Hypersensitivity reaction to omalizumab in the past
* Exceeds limits of dosing table (IgE <30 or 700 IU/ml) or body weight of <30 or > 150kg
* Systemic corticosteroids within the previous month
* Known malignant neoplasm

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-01; Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan Reibman, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omalizumab | Placebo
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: None were on placebo because study had a block randomization of 6.
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab | Placebo | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Measurement in the Reduction of the Effect of Omalizumab on Thymic Stromal Lymphopoietin (TSLP) Using Two Group T-test in Moderate Persistent Asthma
Time Frame: 16 Weeks of Treatment of omalizumab or placebo
Population: Most (n=124) of these patients failed screening criteria and investigator did not move forward
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Measurement in the Reduction of the Effect of Omalizumab on Thymic Stromal Lymphopoietin (TSLP) Using Nonparametric Wilcoxon in sHBEC in Moderate Persistent Asthma
Time Frame: 16 Weeks of Treatment of omalizumab or placebo
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Measurement in the Reduction of the Effect of Omalizumab on IL-33 Gene Expression Using Two Group T-test in Moderate Persistent Asthma
Time Frame: 16 Weeks of Treatment of omalizumab or placebo
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Measurement in the Reduction of the Effect of Omalizumab on IL-33 Gene Expression Using Nonparametric Wilcoxon in sHBEC in Moderate Persistent Asthma
Time Frame: 16 Weeks of Treatment of omalizumab or placebo
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: The Effect of Omalizumab on Changes sHBEC Targets (Gene Expression Array) Compared Using Two-group T-test if Data
Time Frame: 16 Weeks of Treatment of omalizumab or placebo
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Score on Asthma Control Test
Time Frame: 16 Weeks of Treatment of omalizumab or placebo
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Lung Function Measure by Spirometry Test
Time Frame: 16 Weeks of Treatment of omalizumab or placebo
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Measures of Small Airway Dysfunction Using Impulse Oscillometry
Time Frame: 16 Weeks of Treatment of omalizumab or placebo
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: The Effect of Omalizumab on Newly Identified sHBEC Targets (Gene Expression) Analyzed Using Cufflinks.
Time Frame: 16 Weeks of Treatment of omalizumab or placebo
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 0 | 0

10. Other Pre Specified Outcome: The Effect of Omalizumab on Newly Identified sHBEC Targets (Gene Expression) Analyzed Using Gene Analyses
Time Frame: 16 Weeks of Treatment of omalizumab or placebo
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 0 | 0

11. Other Pre Specified Outcome: The Effect of Omalizumab on Gene "Signature" Generation Analyzed Using Gene Analysis Techniques
Time Frame: 16 Weeks of Treatment of omalizumab or placebo
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 60 Months
Description: 0 Patients were on placebo
Arm/Group | Omalizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT02658877/Prot_SAP_000.pdf